CLINICAL TRIAL: NCT02840305
Title: Brain Bases of Visual Perceptionnatural Scenes of Natural Scenes.
Brief Title: Brain Bases of Natural Scenes's Visual Perception of Natural Scenes
Acronym: SCENES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 38RC11.221
Record Dates: First submitted 2016-07-18; First posted 2016-07-21 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2017-01

CONDITIONS: Healthy Volunteer
Keywords: Natural scenes; Brain bases; Visual perception; MRI
MeSH Terms: interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Expérience 1 (Other): Brain bases of spatial frequencies treatment 30 young adults, 20 old adults 20 children between 4 and 6 years, 20 children between 6 and 12 years and 20 young adults
  Interventions: Other: Evaluation of visual function; Other: Magnetic Resonance Imaging
- Expérience 2 (Other): Brain bases of Computer to Film (CtF) analysis 30 young adults, 20 old adults
  Interventions: Other: Evaluation of visual function; Other: Magnetic Resonance Imaging
- Expérience 3 (Other): Part of parahippocampal gyrus in Computer to Film (CtF) analysis 30 young adults, 20 old adults.
  Interventions: Other: Evaluation of visual function; Other: Magnetic Resonance Imaging

INTERVENTIONS:
Other: Evaluation of visual function
Other: Magnetic Resonance Imaging
  Other Names: MRI

SUMMARY:
Using the available data from psychophysics, cellular electrophysiology and functionnal neuroanatomy of visual pathway, current models of visual recognition suppose that the perception of scenes start with a parallel extraction of differents elementary visual characteristics to different spatial frequencies according to a default processing principle named : 'coarse-to-fine'.

According to this principle, the visual scene's analysis would be decomposed in two steps. Fisrt, the fast analysis of the global information borne by low frequency of the scene will provide an overview of the scene's structure and would enable a first perceptive categorisation which would be then refined, approved or denied by the latest analysis of the most local, detailed and precise information, carried by the very high spatial frequency of the scene.

The research carried out since several years is preparing a biologically plausible model and to find brain bases by different imaging techniques among healthy subjects but also patients with a brain lesion and patients with a peripheral lesion.

The main goal of this Magnetic Resonance Imaging study is to find brain bases of natural scenes's visual perception of the natural scenes.

Three studies in Magnetic Resonance Imaging will be conducted, during which subjects will have to categorize pictures of natural scenes filtered in spatial frequencies. The outcome of this study will allow to refine models of visual recognition, most of them based on analysis of spatial frequencies.

ELIGIBILITY:
Inclusion Criteria for young adults :

* Subjet over 18 years and less than 30 years
* Affiliation to a social security
* Free signed consent
* Medical exam done before participation to the study
* Normal or corrected visual acuity

Exclusion Criteria four young adults :

* Counter-argument to MRI
* Pregnant, breast-feeding or parturient women
* Adults non protected or unable to express their consent
* Adults protected
* Important earing or visual disorder
* Neuropsychiatric disorder current or past passée ou présente (exept benign epilepsy)
* Severe affection on a general level (cardiac, respiratory, hematologic, renal, hépatic, cancerous)
* Drug treatment in progress (exept anti-epileptic drug) likely to de modulate brain activity

Inclusion Criteria for old adults :

* Subjet over 50 years
* Affiliation to a social security
* Free signed consent
* Medical exam done before participation to the study
* Normal or corrected visual acuity

Exclusion Criteria four old adults :

* Counter-argument to MRI
* Pregnant, breast-feeding or parturient women
* Adults non protected or unable to express their consent
* Adults protected
* Important earing or visual disorder
* Neuropsychiatric disorder current or past passée ou présente (exept benign epilepsy)
* Severe affection on a general level (cardiac, respiratory, hematologic, renal, hépatic, cancerous)
* Drug treatment in progress (exept anti-epileptic drug) likely to de modulate brain activity

Inclusion Criteria for children :

* Children between 4 and 12 years
* Affiliation to a social security
* Free signed consent
* Medical exam done before participation to the study
* Normal or corrected visual acuity

Exclusion Criteria four children :

* Counter-argument to MRI
* Important earing or visual disorder
* Important development disorder and/or acquisitions identified by parents and/or school teachers
* Neuropsychiatric disorder current or past passée ou présente (exept benign epilepsy)
* Severe affection on a general level (cardiac, respiratory, hematologic, renal, hépatic, cancerous)
* Drug treatment in progress (exept anti-epileptic drug) likely to de modulate brain activity

Min Age: 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 141 (Actual)
Dates: Start 2012-04; Primary Completion 2016-03 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Identify brain bases of natural scenes's visual perception of the natural scenes | About 80 minutes
  Evaluation 1 = Visual tasks Experience 1 : Brain bases of spatial frequencies treatment Experience 2 : Brain bases of Computer to Film (CtF) natural scenes analysis MRI exam Experience 3 : Part of parahippocampal gyrus in Computer to Film (CtF) natural scenes analysis MRI exam About 30 minutes
  Evaluation 2 = Retinotopy : only adults that have shown activations inside occipital cortex during evaluation 1 MRI exam about 50 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre Krainik, Professor, Principal Investigator — Grenoble Hospital University
Locations (1):
- UniversityHospitalGrenoble, La Tronche, France

REFERENCES:
- [Background] Epstein R, Kanwisher N. A cortical representation of the local visual environment. Nature. 1998 Apr 9;392(6676):598-601. doi: 10.1038/33402. PMID 9560155
- [Background] Bar M, Aminoff E, Schacter DL. Scenes unseen: the parahippocampal cortex intrinsically subserves contextual associations, not scenes or places per se. J Neurosci. 2008 Aug 20;28(34):8539-44. doi: 10.1523/JNEUROSCI.0987-08.2008. PMID 18716212
- [Background] Epstein RA, Ward EJ. How reliable are visual context effects in the parahippocampal place area? Cereb Cortex. 2010 Feb;20(2):294-303. doi: 10.1093/cercor/bhp099. Epub 2009 May 20. PMID 19457939
- [Background] Guérin-Dugué, A., & Oliva, A. (1999). Natural images classification from distributions of local dominant orientations, 11th Scandinavian Conference on Image Analysis SCIA'99.
- [Background] Guérin-Dugué, A., & Oliva, A. (2000). Classification of scene photographs from local orientations features. Pattern Recognition Letters, 21, 1135-1140.
- [Background] Hegde J. Time course of visual perception: coarse-to-fine processing and beyond. Prog Neurobiol. 2008 Apr;84(4):405-39. doi: 10.1016/j.pneurobio.2007.09.001. Epub 2007 Sep 29. PMID 17976895
- [Background] Houde O, Pineau A, Leroux G, Poirel N, Perchey G, Lanoe C, Lubin A, Turbelin MR, Rossi S, Simon G, Delcroix N, Lamberton F, Vigneau M, Wisniewski G, Vicet JR, Mazoyer B. Functional magnetic resonance imaging study of Piaget's conservation-of-number task in preschool and school-age children: a neo-Piagetian approach. J Exp Child Psychol. 2011 Nov;110(3):332-46. doi: 10.1016/j.jecp.2011.04.008. Epub 2011 Jun 1. PMID 21636095
- [Background] Hérault, J., Oliva, A., & Guérin-Dugué, A. (1997). Scene categorisation by curvilinear component analysis of low frequency spectra. Paper presented at the IANN'97, Bruges
- [Background] Hubel DH, Wiesel TN. Ferrier lecture. Functional architecture of macaque monkey visual cortex. Proc R Soc Lond B Biol Sci. 1977 Jul 28;198(1130):1-59. doi: 10.1098/rspb.1977.0085. No abstract available. PMID 20635
- [Background] Hughes HC, Nozawa G, Kitterle F. Global precedence, spatial frequency channels, and the statistics of natural images. J Cogn Neurosci. 1996 Summer;8(3):197-230. doi: 10.1162/jocn.1996.8.3.197. PMID 23968149
- [Background] Kimchi R. Primacy of wholistic processing and global/local paradigm: a critical review. Psychol Bull. 1992 Jul;112(1):24-38. doi: 10.1037/0033-2909.112.1.24. PMID 1529037
- [Background] Lamb MR, Yund EW. The role of spatial frequency in the processing of hierarchically organized stimuli. Percept Psychophys. 1993 Dec;54(6):773-84. doi: 10.3758/bf03211802. PMID 8134247
- [Background] Lux S, Marshall JC, Thimm M, Fink GR. Differential processing of hierarchical visual stimuli in young and older healthy adults: implications for pathology. Cortex. 2008 Jan;44(1):21-8. doi: 10.1016/j.cortex.2005.08.001. Epub 2007 Nov 17. PMID 18387528
- [Background] Monoyer, F. (1875). Echelle typographique pour la détermination de l'acuité visuelle. (Acad. des Sciences, Comptes rendus). Gaz. Méd. De Paris, 80, 113.
- [Background] Musel B, Chauvin A, Guyader N, Chokron S, Peyrin C. Is coarse-to-fine strategy sensitive to normal aging? PLoS One. 2012;7(6):e38493. doi: 10.1371/journal.pone.0038493. Epub 2012 Jun 4. PMID 22675568
- [Background] Navon, D. (1977). Forest before trees: the precedence of global features in visual perception. Cognitive Psychology, 9, 353-383.
- [Background] Oken BS, Kishiyama SS, Kaye JA, Jones DE. Age-related differences in global-local processing: stability of laterality differences but disproportionate impairment in global processing. J Geriatr Psychiatry Neurol. 1999 Summer;12(2):76-81. doi: 10.1177/089198879901200207. PMID 10483929
- [Background] Oliva, A. (1995). Perception de scènes: Traitement fréquentiel du signal visuel aspects psychophysiques et neurophysiologiques. Institut National Polytechnique, Grenoble.
- [Background] Oliva A, Schyns PG. Coarse blobs or fine edges? Evidence that information diagnosticity changes the perception of complex visual stimuli. Cogn Psychol. 1997 Oct;34(1):72-107. doi: 10.1006/cogp.1997.0667. PMID 9325010
- [Background] Park S, Brady TF, Greene MR, Oliva A. Disentangling scene content from spatial boundary: complementary roles for the parahippocampal place area and lateral occipital complex in representing real-world scenes. J Neurosci. 2011 Jan 26;31(4):1333-40. doi: 10.1523/JNEUROSCI.3885-10.2011. PMID 21273418
- [Background] Pelli, D. G., Robson, J. G., & Wilkins, A. J. (1988). The design of a new letter chart for measuring contrast sensitivity. Clinical Vision Sciences, 2(3), 187-199.
- [Background] Peyrin C, Baciu M, Segebarth C, Marendaz C. Cerebral regions and hemispheric specialization for processing spatial frequencies during natural scene recognition. An event-related fMRI study. Neuroimage. 2004 Oct;23(2):698-707. doi: 10.1016/j.neuroimage.2004.06.020. PMID 15488419
- [Background] Peyrin C, Chauvin A, Chokron S, Marendaz C. Hemispheric specialization for spatial frequency processing in the analysis of natural scenes. Brain Cogn. 2003 Nov;53(2):278-82. doi: 10.1016/s0278-2626(03)00126-x. PMID 14607164
- [Background] Peyrin C, Chokron S, Guyader N, Gout O, Moret J, Marendaz C. Neural correlates of spatial frequency processing: A neuropsychological approach. Brain Res. 2006 Feb 16;1073-1074:1-10. doi: 10.1016/j.brainres.2005.12.051. Epub 2006 Jan 27. PMID 16443206
- [Background] Peyrin C, Mermillod M, Chokron S, Marendaz C. Effect of temporal constraints on hemispheric asymmetries during spatial frequency processing. Brain Cogn. 2006 Dec;62(3):214-20. doi: 10.1016/j.bandc.2006.05.005. Epub 2006 Jul 11. PMID 16837115
- [Background] Peyrin C, Michel CM, Schwartz S, Thut G, Seghier M, Landis T, Marendaz C, Vuilleumier P. The neural substrates and timing of top-down processes during coarse-to-fine categorization of visual scenes: a combined fMRI and ERP study. J Cogn Neurosci. 2010 Dec;22(12):2768-80. doi: 10.1162/jocn.2010.21424. PMID 20044901
- [Background] Peyrin C, Schwartz S, Seghier M, Michel C, Landis T, Vuilleumier P. Hemispheric specialization of human inferior temporal cortex during coarse-to-fine and fine-to-coarse analysis of natural visual scenes. Neuroimage. 2005 Nov 1;28(2):464-73. doi: 10.1016/j.neuroimage.2005.06.006. Epub 2005 Jul 1. PMID 15993630
- [Background] Poirel N, Mellet E, Houde O, Pineau A. First came the trees, then the forest: developmental changes during childhood in the processing of visual local-global patterns according to the meaningfulness of the stimuli. Dev Psychol. 2008 Jan;44(1):245-53. doi: 10.1037/0012-1649.44.1.245. PMID 18194023
- [Background] Poirel N, Simon G, Cassotti M, Leroux G, Perchey G, Lanoe C, Lubin A, Turbelin MR, Rossi S, Pineau A, Houde O. The shift from local to global visual processing in 6-year-old children is associated with grey matter loss. PLoS One. 2011;6(6):e20879. doi: 10.1371/journal.pone.0020879. Epub 2011 Jun 8. PMID 21687636
- [Background] Shulman GL, Sullivan MA, Gish K, Sakoda WJ. The role of spatial-frequency channels in the perception of local and global structure. Perception. 1986;15(3):259-73. doi: 10.1068/p150259. PMID 3797200
- [Background] Shulman GL, Wilson J. Spatial frequency and selective attention to local and global information. Perception. 1987;16(1):89-101. doi: 10.1068/p160089. PMID 3671045
- [Background] Schyns, P. G., & Oliva, A. (1994). From blobs to boundary edges: Evidence for time- and spatial-scale-dependant scene recognition. American Psychological Society, 5, 195-200.
- [Background] Schyns PG, Oliva A. Flexible, diagnosticity-driven, rather than fixed, perceptually determined scale selection in scene and face recognition. Perception. 1997;26(8):1027-38. doi: 10.1068/p261027. PMID 9509161
- [Background] Schyns PG, Oliva A. Dr. Angry and Mr. Smile: when categorization flexibly modifies the perception of faces in rapid visual presentations. Cognition. 1999 Jan 1;69(3):243-65. doi: 10.1016/s0010-0277(98)00069-9. PMID 10193048
- [Background] Staudinger MR, Fink GR, Mackay CE, Lux S. Gestalt perception and the decline of global precedence in older subjects. Cortex. 2011 Jul-Aug;47(7):854-62. doi: 10.1016/j.cortex.2010.08.001. Epub 2010 Aug 11. PMID 20828678
- [Background] Van Essen, D. C., & DeYoe, E. A. (1995). Concurrent processing in the primate visual cortex. In M. Gazzaniga (Ed.), The cognitive Neurosciences (pp. 383-400). Cambridge: Bradford Book.
- [Background] Vasseur F, Delon-Martin C, Bordier C, Warnking J, Lamalle L, Segebarth C, Dojat M. fMRI retinotopic mapping at 3 T: benefits gained from correcting the spatial distortions due to static field inhomogeneity. J Vis. 2010 Oct 26;10(12):30. doi: 10.1167/10.12.30. PMID 21047762
- [Background] Warnking J, Dojat M, Guerin-Dugue A, Delon-Martin C, Olympieff S, Richard N, Chehikian A, Segebarth C. fMRI retinotopic mapping--step by step. Neuroimage. 2002 Dec;17(4):1665-83. doi: 10.1006/nimg.2002.1304. PMID 12498741